CLINICAL TRIAL: NCT06662812
Title: Disease Characteristics and Treatment Patterns of Patients With Sickle Cell Disease in Globin Research Network for Data and Discovery (GRNDaD) Registry
Brief Title: Characteristics and Treatment Patterns of Patients With Sickle Cell Disease in Globin Research Network for Data and Discovery Registry
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CSEG101AUS19
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- GRNDaD Cohort: Patients with sickle cell disease (SCD) who were included in the GRNDaD registry and received a disease modifying therapy (DMT).

SUMMARY:
This was a retrospective observational cohort study. This study was a secondary analysis of individuals with sickle cell disease (SCD) enrolled in the GRNDaD registry.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of SCD.
* Signed consent to participate in GRNDaD registry.

Exclusion criteria:

• None identified at this time.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 1665 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Number of Patients in the Globin Research Network for Data and Discovery (GRNDaD) Registry who Received a Disease Modifying Therapy (DMT) | Up to 2 years
  DMTs included: hydroxyurea, voxelotor, crizanlizumab, l-glutamine, and chronic red cell transfusion.

SECONDARY OUTCOMES:
Number of Patients in the Globin Research Network for Data and Discovery (GRNDaD) Registry Using Hydroxyurea Categorized by Gender | Up to 2 years
Number of Patients in the GRNDaD Registry Using Hydroxyurea Categorized by Genotype | Up to 2 years
Number of Patients in the GRNDaD Registry Using Hydroxyurea Categorized by Age | Up to 2 years
Number of Patients in the GRNDaD Registry Using Voxelotor Categorized by Gender | Up to 2 years
Number of Patients in the GRNDaD Registry Using Voxelotor Categorized by Genotype | Up to 2 years
Number of Patients in the GRNDaD Registry Using Voxelotor Categorized by Age | Up to 2 years
Number of Patients in the GRNDaD Registry Using Crizanlizumab Categorized by Gender | Up to 2 years
Number of Patients in the GRNDaD Registry Using Crizanlizumab Categorized by Genotype | Up to 2 years
Number of Patients in the GRNDaD Registry Using Crizanlizumab Categorized by Age | Up to 2 years
Number of Patients in the GRNDaD Registry Using L-glutamine Categorized by Gender | Up to 2 years
Number of Patients in the GRNDaD Registry Using L-glutamine Categorized by Genotype | Up to 2 years
Number of Patients in the GRNDaD Registry Using L-glutamine Categorized by Age | Up to 2 years
Number of Patients in the GRNDaD Registry Using Chronic Transfusion Categorized by Gender | Up to 2 years
Number of Patients in the GRNDaD Registry Using Chronic Transfusion Categorized by Genotype | Up to 2 years
Number of Patients in the GRNDaD Registry Using Chronic Transfusion Categorized by Age | Up to 2 years
Number of Hospital Admissions Categorized by Age | Up to 2 years
Mean Number of Hospital Admissions | Up to 2 years
Number of Emergency Department Visits Categorized by Age | Up to 2 years
Mean Number of Emergency Department Visits | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States